CLINICAL TRIAL: NCT03817333
Title: The Mixed Phenotype of Asthma and COPD: the Overlap Syndrome: A Comparison of Asthma Outcomes in Smoking vs Non-smoking Patients With an Incomplete Reversibility of Airway Obstruction (IRAO)
Brief Title: The Mixed Phenotype of Asthma and COPD: the Overlap Syndrome
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: CÉR21047
Record Dates: First submitted 2016-01-13; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Asthma; COPD
Keywords: phenotype; inflammation; pulmonary function; comorbidities
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACOS smoking history >20 pack-years: Subjects with asthma-COPD overlap syndrome
- IRAO smoking history <5 pack-years: Subjects with an incomplete reversibility of airway obstruction

SUMMARY:
RATIONALE:

In asthmatic subjects, smoking can lead to several changes in disease characterictics. in smokers of more than 20 pack-years, chronic obstructive pulmonary disease (COPD) can be associated with asthma, also called asthma-COPD overlap syndrome (ACOS). Increasing data support the concept that ACOS is a clinical entity. However, this should be further studied in order to better target therapy.

AIM:

The objective of this study is to evaluate the comparative features of ACOS

METHODS:

This will be a descriptive study comparing the features of the ACOS with the features of asthmatic subjects with an incomplete reversibility of airway obstruction (IRAO).The study will be done over 1 or 2 visits (within a week interval), according to subjects' availability. The visit will include completion of different questionnaires (asthma control asthma quality of life, medical history, exacerbations, etc.), a thoracic examination, allergy skin-prick tests, spirometry and bronchodilator response, lung volumes and compliance measurements, exhaled nitric oxide measurement, blood sampling and a sputum induction.

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS

1. Subjects aged 45 years and older.
2. Free of any other respiratory condition, except for asthma and/or COPD, which may interfere with the tests.
3. Asthma that requires a baseline treatment with inhaled corticosteroids and/or additional asthma medication.
4. Free of respiratory infection in the 4 weeks preceding the study.
5. No changes in the asthma and COPD-related medications in the 4 weeks preceding the study.
6. If female, not pregnant (or lactating).
7. Able to adhere to study procedures.
8. Able and willing to provide written informed consent to participate in the study, in accordance with international conference on harmonization (ICH) good clinical practice (GCP) requirements.

ACOS SUBJECTS

1. Smokers or ex-smokers of at least 20 pack-years. 2. With an IRAO (see definitions section). IRAO SUBJECTS

1. Long-life non-smokers or ex-smokers defined as someone who smoked less than 5 pack-years and who completely stopped smoking for at least 12 months before inclusion in the study.
2. With an IRAO.

Exclusion Criteria:

* ALL SUBJECTS

  1. With COPD without a past diagnosis of asthma.
  2. Unstable respiratory or non-respiratory condition.
  3. Any active chronic inflammatory disease.
  4. Any evidence of malignancy (active and/or treated) within the previous 5 years.
  5. Any significant concomitant illness or injury that would interfere with the subject's participation in the study.
  6. Any history of bronchial thermoplasty. IRAO SUBJECTS

  <!-- -->

  1. Use of any nicotine containing product within 1 year prior to study entry or a smoking history of > 5 pack-years.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic subjects will be recruited from the asthma outpatient clinic, from participation to past research studies, or from advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Total asthma control questionnaire (ACQ) score | Baseline
  Measurement of asthma control using a 0-6 scale. The questionnaire includes 6 questions. Total score is the mean of the scores from all questions. Total score ranges from 0 to 6. A lower score is better.

SECONDARY OUTCOMES:
Spirometry results | Baseline
  Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC
Sputum eosinophil percentage | Baseline
  Percentage of sputum eosinophils
Concentration of Blood biomarkers | Baseline
  alpha 1 antitrypsine, C-reactive protein (CRP), fibrinogen
Asthma quality of life questionnaire (AQLQ) score | Baseline
  Measurement of asthma quality of life using the Mini asthma quality of life questionnaire. It is a 7-point scale questionnaire (where 1 is greatest impairment and 7 is least impairment) containing 15 uqestions divided into 4 domains : symptoms (5 items), activity limitation (4 items), emotional function (3 items), and exposure to environmental stimuli (3 items). during the last 2 weeks. The overall score is the mean of all the responses. Each domain score is calculated from the mean of the items that relate to it.
Number of patients with comorbidities | Baseline
  gastro-oesophageal reflux disease (GERD), obstructive sleep apnea (OSA), anxiety, depression
Number of asthma exacerbations in the previous year | Baseline
  emergency room (ER) visits, hospitalizations, oral corticosteroids treatment, unscheduled medical visits
Change from baseline total Asthma Control Questionnaire (ACQ) score at one-year follow-up | Baseline to one-year follow-up
  Measurement of asthma control using a 0-6 scale. The questionnaire includes 6 questions. Total score is the mean of the scores from all questions. Total score ranges from 0 to 6. A lower score is better.
Change from baseline number of exacerbations at one-year follow-up | Baseline to one-year follow-up
  emergency room (ER) visits, hospitalizations, oral corticosteroids treatment, unscheduled medical visits

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada